CLINICAL TRIAL: NCT06280963
Title: Posterior Innominate Mobilization Versus Muscle Energy Technique on Lumbopelvic Angles in Sacroiliac Joint Dysfunction
Acronym: MET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Yousry Rashwan Hefny (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Yousry Rashwan Hefny, Senior Physical Therapist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 012/005532
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Sacroiliac Joint Dysfunction
Keywords: lumbopelvic angles; muscle energy technique; sacroiliac joint dysfunction; posterior innominate mobilization

STUDY DESIGN:
Intervention Model Description: group one will receive muscle energy technique group two will receive posterior innominate mobilization group three will receive conventional treatment ( TENS , US , stertching exercises and strenghening exercises )
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- muscle energy technique arm (Experimental): this arm will receive muscle energy technique
  Interventions: Behavioral: muscle energy technique
- posterior innominate mobilization arm (Experimental): this arm will receive posterior innominate mobilization
  Interventions: Behavioral: posterior innominate mobilization
- control arm (Placebo Comparator): this arm will receive conventional treatment
  Interventions: Behavioral: conventional treatment

INTERVENTIONS:
Behavioral: muscle energy technique — in muscle energy technique, the target is gluteus maximus muscle ( hip extension ) and repeat the method from three to five times .
  Arms: muscle energy technique arm
Behavioral: posterior innominate mobilization — in posterior innominate mobilization ( grade 3 mobilization ) , frequency of mobilizations is 30 oscillations , 3 sets per session ( every set has 30 oscillations )
  Arms: posterior innominate mobilization arm
Behavioral: conventional treatment — conventional treatment include
  * TENS ( 45 minutes of conventional TENS )
  * Ultrasound (pulsed mode 1:1 ,5 min .1.5W/cm2 )
  * Stretching exercises ( hamstrings ,hip flexors and hip adductors)
  * Strengthening exercises (lower abdomen and glutes muscles )
  * Lumpopelvic stabilization exercise
  Other Names: placebo treatment
  Arms: control arm

SUMMARY:
the goal of this clinical trial study is to compare between posterior innominate mobilization and muscle energy techniqueon lumbopelvic angles in sacroiliac joint dysfunction patients.

the main questions they aim to answer are

1. are there statistical significant effects of posterior innominate mobilization versus muscle energy technique on lumbopelvic angles in sacroiliac joint dysfunction patients ?
2. are there statistical significant effects of posterior innominate mobilization versus muscle energy technique on pain intensity level in sacroiliac joint dysfunction patients ?

   * purpose of the study is to measure the effect of muscle energy technique versus posterior innominate mobilization on lumbopelvic angles in sacroiliac joint dysfunction

DETAILED DESCRIPTION:
Sacroiliac joint dysfunction ( SIJ ) refers to a state of altered biomechanics of the SIJ. The sacrum does not exhibit muscle motion with respect to the ilium and SIJs are slackened only during pregnancy. Excessive or restricted motion may affect extra-articular structures surrounding the SIJs (such as the sacrotuberous, sacrospinus, and/or iliolumbar ligaments) and results in pain.

Sacroiliac (SI) joint dysfunction is a common cause of low back pain and accurate diagnosis can be challenging. A complete history and physical examination are critical in differentiating other diagnosis that may have similar signs and symptoms. Positive response to at least three physical provocation tests suggest sacroiliac joint dysfunction.

Muscle Energy Technique (MET) is an active technique in which the patient is also an active participant. MET is based on the concepts of Autogenic Inhibition and Reciprocal Inhibition. If a sub-maximal contraction of the muscle is followed by stretching of the same muscle it is known as Autogenic Inhibition MET, and if a submaximal contraction of a muscle is followed by stretching of the opposite muscle then this is known as Reciprocal Inhibition MET.

SIJ mobilization is a method of physical therapy. The advantages of the SIJ mobilization are reported in many aspects, such as decrease of LBP, decrease lumbar spinal stress by restoring normal function of innominate, promote pelvic symmetry, correct the sacroiliac joint dysfunction and relax surrounding muscles of the SIJ delimitations are

* Patients suffering from SIJ dysfunction with age between 25 and 45
* Patients with pain in gluteal region and around SIJ.
* Patients testing positive in at least 3 of the following test:

  1. Gaenslen's test
  2. . Standing forward bending test
  3. . Sacroiliac distraction test
  4. . Sacroiliac compression test
  5. . Patrick and fabric test
* Patients with visual analogue scale more than 3.\ lumbopelvic angles are four spinopelvic parameters which are

  1. Lumbar lordotic angle: The angle between the upper plate of the first lumbar and first sacral vertebral bodies .Mean value of lumber lordotic angle is 65.4
  2. Pelvic incidence: Through the intersection of the line perpendicular to the sacral plate at its midpoint and the line connecting the point to the middle axis of the femoral heads .

     Mean value of pelvic incidence is 51.50
  3. Pelvic tilt: Assessed by the intersection of the lines that cross the midpoint of both centers of the femoral heads and the mid-point of the sacral plateau with the line perpendicular to the ground. Mean value of pelvic tilt is 12.32
  4. Sacral slope: Through the intersection of lines parallel to the sacral plateau and parallel to the ground . Mean value of sacral slope is 39.17 * CorelDraw: is a family of software programs used for editing vector graphics, illustration and design. It is used in health care to measure spinopelvic angles after taking photos of them from their x-rays on mobile.

inclusion criteria : Subjects with sacroiliac joint dysfunction of both sexes with all the following criteria:

* Internal torsion of ilium on sacrum in sacroiliac joint dysfunction patients
* Normal weight - BMI greater than or equal to 18.5 to 24.9 kg/m^2
* Patients with age from 25 to 45
* Patients with VAS more than 3
* Pain around SIJ and groin area
* Patients testing positive at least 3 of six SIJ pain provocation tests (Gaenslen's test, Distraction test, Compression test, Thigh thrust test, Sacral thrust test, Patrick and fabric test)

Exclusion criteria: Patients will be excluded if they exhibited any of the following:

* Underlying neuro defects in leg
* Sacroiliitis
* Spondylolisthesis
* prediagnosed disease of central or peripheral nervous system
* Current pregnancy
* Rheumatological disease
* History of major surgery of lower extremity or spine
* Osteoporosis
* Recent injection of corticosteroids in SIJ

evaluation instruments :

1. visual analogue scale (VAS) : a tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount the amount of pain he or she feels . It will be used to assess current level of sacroiliac joint pain. Once subjects reported a pain level more than 3 on the visual analog scale [VAS], it will be included in the study. It has a Moderate to good reliability in patients with chronic musculoskeletal pain
2. X-rays are form of electromagnetic radiation, similar to visible light. Unlike light, however, x-rays have higher energy and can pass through most objects, including the body. Medical x-rays are used to generate images of tissues and structures inside the body. If x-rays traveling through the body also pass through an x-ray detector on the other side of the patient, an image will be formed that represents the "shadows" formed by the objects inside of the body. One type of x-ray detector is photographic film, but there are many other types of detectors that are used to produce digital images. The x-ray images that result from this process are called radiographs.
3. CorelDraw for measurement of lumbopelvic angels. It is used in health care to measure spinopelvic angles after taking photos of them from their x-rays on mobile.

After taking lumbopelvic x-ray from lateral view for all subjects from standing position . Put each X ray on lighting unit and take a photo by mobile camera. Put all soft copies of X ray pictures on a computer and measure the spinopelvic angels (sacral slope, lumber lordosis, pelvic incidence and pelvic tilt) by using CorelDraw graphic suits.

treatment tools and procedures :

1. muscle energy technique : In this study post isometric relaxation on gluteus maximus will be used:-

   * Patient position: side lying with lower most leg extended and upper most leg flexed at hip and knee joint and held by therapist hand and his pelvis.
   * Therapist position: stand in front of the patient with wide base of support one hand on PSIS and other hand hold the femur of the patient.
   * Order: ask the patient to push his femur toward the therapist hand ( hip extension for glutes maximus muscle ) and hold for five to seven seconds, then relax and the therapist will get a new barrier and repeat this method for three to five times
2. Posterior innominate mobilization

   * Patient position: side lying with lower most leg extended and upper most leg flexed at hip and knee joints.
   * Therapist position: stand in front of the patient one hand on anterior superior iliac spine( ASIS) and his another forearm on the buttock.
   * Procedure: pull ASIS backward (grade 3 mobilization). Frequency of mobilization: 30 oscillations , 3 sets per session ( every set has 30 oscillations )

ELIGIBILITY:
Inclusion Criteria:

* Internal torsion of ilium on sacrum in sacroiliac joint dysfunction patients
* Normal weight - BMI greater than or equal to 18.5 to 24.9 kg/m^2
* Patients with age from 25 to 45
* Patients with VAS more than 3
* Pain around SIJ and groin area
* Patients testing positive at least 3 of six SIJ pain provocation tests (Ganesen's test, Distraction test, Compression test, Thigh thrust test, Sacral thrust test, Patrick and fabric test)

Exclusion Criteria:

* Underlying neuro defects in leg
* Sacroiliitis
* Spondylolisthesis
* Pre diagnosed disease of central or peripheral nervous system
* Current pregnancy
* Rheumatological disease
* History of major surgery of lower extremity or spine
* Osteoporosis
* Recent injection of corticosteroids in SIJ

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-03 (Estimated)

PRIMARY OUTCOMES:
lumbopelvic angles | 2 days
  measurement of lumbopelvic angle ( pelvic incidence , sacral slope , lumbar lordosis and pelvic tilt

SECONDARY OUTCOMES:
pain intensity | about 2 days
  measurement of pain intensity by visual analogue scale It will be used to assess current level of sacroiliac joint pain. Once subjects reported a pain level more than 3 on the visual analog scale [VAS], it will be included in the study

CONTACTS AND LOCATIONS:
Overall Officials: Haytham M Elhafez, Study Director — faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiapour A, Joukar A, Elgafy H, Erbulut DU, Agarwal AK, Goel VK. Biomechanics of the Sacroiliac Joint: Anatomy, Function, Biomechanics, Sexual Dimorphism, and Causes of Pain. Int J Spine Surg. 2020 Feb 10;14(Suppl 1):3-13. doi: 10.14444/6077. eCollection 2020 Feb. PMID 32123652
- [Background] Nejati P, Safarcherati A, Karimi F. Effectiveness of Exercise Therapy and Manipulation on Sacroiliac Joint Dysfunction: A Randomized Controlled Trial. Pain Physician. 2019 Jan;22(1):53-61. PMID 30700068
- [Result] Dydyk, A. M., Forro, S. D., & Hanna, A. (2020). Sacroiliac joint injury. StatPearls Publishing, Treasure Island (FL), 04 Jun 2020 PMID: 32491804
- See also: Effects of mobilization treatment on sacroiliac joint dysfunction syndrome — https://doi.org/10.1590/1806-9282.20210436